CLINICAL TRIAL: NCT01547546
Title: An Open-label, Phase I, Dose-escalation Study Evaluating the Safety and Tolerability of GDC-0084 Administered to Patients With Progressive or Recurrent High-grade Glioma
Brief Title: A Study of GDC-0084 in Patients With Progressive or Recurrent High-Grade Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO28070; 2011-004479-35 (EudraCT Number)
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Glioblastoma, Glioma
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — GDC-0084

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: GDC-0084

INTERVENTIONS:
Drug: GDC-0084 — Multiple doses

SUMMARY:
This open-label, multicenter, Phase I, dose-escalating study will evaluate the safety and tolerability, pharmacokinetics, pharmacodynamics and efficacy of GDC-0084 in patients with progressive or recurrent high-grade glioma. Stage 1 is the dose escalation part of the study. Stage 2, patients will receive GDC-0084 at a recommended dose for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Interval of at least 12 weeks from completion of adjuvant radiotherapy for gliomas to study entry
* Karnofsky Performance Status of >/= 70 at screening
* Confirmed measurable disease per RANO
* Adequate hematologic and organ function

Patients enrolled in Stage 1:

* Histologically documented recurrent or progressive high-grade gliomas (WHO Grade III-IV)
* Prior treatment with at least one regimen for gliomas (radiotherapy with or without chemotherapy for Grade III gliomas and radiotherapy with chemotherapy for Grade IV gliomas) and/or not considered to be a candidate for regimens known to provide clinical benefit

Patients enrolled in Stage 2:

* Histologically documented recurrent or progressive glioblastoma (WHO Grade IV gliomas)
* Prior treatment with one or two regimens for glioblastoma (with the initial regimen consisting of radiotherapy with chemotherapy)

Exclusion Criteria:

* Treatment with anti-tumor therapy (approved or experimental) within 4 weeks prior to initiation of study drug
* Requirement for anticoagulants such as warfarin or any other warfarin-derivative anticoagulants; low-molecular-weight heparin is permitted
* Any contraindication to MRI examination
* Evidence of Grade >/= 1 intracranial hemorrhage
* Active congestive heart failure or ventricular arrhythmia requiring medication
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse or cirrhosis
* Unresolved toxicity from prior therapy with the exception of lymphopenia (for patients with prior temozolomide) and alopecia
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | approximately 2 years
Maximum tolerated dose (MTD) | approximately 1 year

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the concentration-time curve | Pre- and post-dose Days 1, 8, 15, 22 and 29 Cycle 1, Day 1 every following Cycle until 30 days after the last dose of study drug
Best overall response rate, tumor assessments according to Response Assessment in Neuro-Oncology (RANO) | approximately 2 years
Duration of response | approximately 2 years
Progression-free survival | approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (4):
- United States (3):
  - Los Angeles, California
  - Boston, Massachusetts
  - Houston, Texas
- Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Ellingson BM, Yao J, Raymond C, Nathanson DA, Chakhoyan A, Simpson J, Garner JS, Olivero AG, Mueller LU, Rodon J, Gerstner E, Cloughesy TF, Wen PY. Multiparametric MR-PET Imaging Predicts Pharmacokinetics and Clinical Response to GDC-0084 in Patients with Recurrent High-Grade Glioma. Clin Cancer Res. 2020 Jul 1;26(13):3135-3144. doi: 10.1158/1078-0432.CCR-19-3817. Epub 2020 Apr 8. PMID 32269051
- [Derived] Wen PY, Cloughesy TF, Olivero AG, Morrissey KM, Wilson TR, Lu X, Mueller LU, Coimbra AF, Ellingson BM, Gerstner E, Lee EQ, Rodon J. First-in-Human Phase I Study to Evaluate the Brain-Penetrant PI3K/mTOR Inhibitor GDC-0084 in Patients with Progressive or Recurrent High-Grade Glioma. Clin Cancer Res. 2020 Apr 15;26(8):1820-1828. doi: 10.1158/1078-0432.CCR-19-2808. Epub 2020 Jan 14. PMID 31937616